| CT.gov RISE Statistical Analysis Plan 210628 |
|---|
| Research and Innovation to Stop E-cigarette/Vaping in Young Adults Statistical Analysis Plan |
| ID # GR120236<br>NCT ID: Not yet assigned |
| June 28, 2021 |

Descriptive statistics will be used to characterize the sample randomized to each of the four (2x2) arms. A logistic regression model will be used to estimate the main effect of each factor while controlling for the other on the primary outcome - self-reported 7-day point prevalence abstinence (yes/no) assessed at 3 months. Consistent with the MOST design, each factor will be tested against the null using an alpha of 0.1 as a balance of the potential for type I and type II at this phase of intervention development. A second logistic regression model will examine the two-way interaction between the factors as a secondary analysis. The primary analysis will consider all those lost to follow up as non-abstinent; sensitivity analyses will use multiple imputation for the missing values.